CLINICAL TRIAL: NCT03667430
Title: Tolerability and Feasibility Evaluation of a Food Additive Based on Porous Silica Compounds for Future Weight Loss and Prevention of Obesity Related Co-morbidities
Brief Title: Safety Evaluation of Porous Silica in Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Sigrid Therapeutics AB, Sweden (Industry); Stockholm University (Other)
Responsible Party: Principal Investigator, Pernilla Danielsson, Principal Investigator, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Sigrid1
Record Dates: First submitted 2018-08-23; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Safety Issues
MeSH Terms: interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal weight subjects (Experimental): Healthy normal weight (BMI 20-25) men 18-35 year. Intervention: The participants will take placebo or silica powder with specified doses administrated in vials and with instructions to mix with water as; Placebo (microcrystalline cellulose) day 1-5 Porous silica 1gx3 daily for day 6-9 Porous silica 2gx3 daily for day 10-14 Porous silica 3gx3 daily for day 15-21 Total study time 21 days
  Interventions: Dietary Supplement: Porous silica; Dietary Supplement: Placebo (microcrystalline cellulose)
- Subjects with obesity (Experimental): Obese otherwise healthy men (BMI 30-45) 18-35 year Intervention: The participants will take placebo or silica powder with specified doses administrated in vials and with instructions to mix with water as; Placebo (microcrystalline cellulose) day 1-5 Porous silica 1gx3 daily for day 6-9 Porous silica 2gx3 daily for day 10-14 Porous silica 3gx3 daily for day 15-21 The dose of Silica 3gx3 for additional 10 weeks Total study time 84 days
  Interventions: Dietary Supplement: Porous silica; Dietary Supplement: Placebo (microcrystalline cellulose)

INTERVENTIONS:
Dietary Supplement: Porous silica — The particle is rod shaped and approximately 1-3 x 0.4-0.5 micrometers with pore sizes in the range of 70-130 Ångström or 7-13 nanometer.
Dietary Supplement: Placebo (microcrystalline cellulose) — All participants starts with five days placebo run in period

SUMMARY:
The aim of the present study was to determine whether oral dosing, up to 9 grams/day, of porous silica administered as a food additive can be used safely in normal weight and obese male humans, without significant side effects on gastrointestinal function, bowel emptying habits, and biomarkers.

DETAILED DESCRIPTION:
This single blinded safety study will consist of two study arms and include 10 males each (18-35 years). One arm will include participants with normal weight and one with obesity. After a placebo run-in period, all subjects will be given porous silica three times daily, with increasing dose up to 9 grams/day (Phase 1). Subjects with obesity continued the study with highest dose for additional 10 weeks (Phase 2).

The participants will have weekly contacts during with the representative for the study (PI or other research staff). Clinical examinations, and blood sampling will be performed day 1, 7, 14, and 21. Faeces and morning urinary sampling day 1, and 21. Information regarding eating habits, sleep patterns, living conditions and gastrointestinal health were obtained from written forms and orally. If gastrointestinal adverse events would occur after increased dosage, the study staff will adapt the dosage protocol to facilitate adherence.

ELIGIBILITY:
Inclusion Criteria:

Group - Normal weight subjects

* Age 18-35
* BMI 20-25

Group - Subject with obesity

* Age 18-35
* BMI 30-45

Exclusion Criteria:

* Chronic somatic diseases that may affect metabolic and/or intestinal function (e.g. diabetes, hypertension, dyslipidemia, Irritable Bowel Disease, gluten intolerance, pancreatic dysfunction, other causes of malabsorption, neoplastic disease,)
* Allergies with previous anaphylactic reactions
* Previous abdominal surgery
* Current or history of eating disorders
* Extreme or unusual diets such as Low Carb High Fat and vegetarian diets for the last year
* Psychiatric disorders (e.g. schizophrenia, and other diagnoses that may influence compliance)
* Drug or alcohol abuse
* Continuous oral pharmacological treatment and other types of pharmacological treatment that may influence the study
* Other conditions which the investigator considers could negatively affect the outcome of the study or study compliance

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-02-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | From start of intervention up to 12 weeks
  According to MedDRA SOC.

SECONDARY OUTCOMES:
Number of participants with affected gastrointestinal function | From start of intervention up to 12 weeks
  Evaluates by 5 graded questions of gastrointestinal habits and discomfort
Presence of fecal abnormalities | From start of intervention up to 12 weeks
  Tests of Hemoglobin, calprotectin and elastase in feces
Change in nutrition status | From start of intervention up to 12 weeks
  Vitamin and trace elements levels measured in blood
Change in lipid profile | From start of intervention up to 12 weeks
  Triglycerides, total cholesterol, high density lipoprotein cholesterol, low density lipoprotein cholesterol in blood
Change in glucose metabolism | From start of intervention up to 12 weeks
  Fasting glucose, insulin and hemoglobin A1c in blood
Change in liver status | From start of intervention up to 12 weeks
  Alanine aminotransferase and aspartate aminotransferase in blood
Change in renal status measured by creatinine | From start of intervention up to 12 weeks
  Creatinine in blood
Change in renal status measured by glomerular filtration rate | From start of intervention up to 12 weeks
  Glomerular filtration rate in blood
Change in renal status measured by cystatin C | From start of intervention up to 12 weeks
  Cystatin C in blood
Change in concentration of silica | From start of intervention up to 12 weeks
  Urine sample
Change in systemic inflammation status | From start of intervention up to 12 weeks
  C-reactive protein in blood
Change in blood pressure | From start of intervention up to 12 weeks
  Diastolic and systolic blood pressure
Body weight | From start of intervention up to 12 weeks
  Weight (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Danielsson, PhD, Principal Investigator — Karolinska Institutet